CLINICAL TRIAL: NCT05041582
Title: Combining SSRIs and TDCS to Enhance Motor Recovery After Stroke
Brief Title: SSRIs and TDCS Enhance Post-stroke Motor Recovery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chih-Wei Tang (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Chih-Wei Tang, Chief, Stroke Center, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Co-STARS
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Motor
Keywords: stroke, motor recovery, transcranial direct current stimulation, selective serotonin reuptake inhibitors
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Citalopram; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real tDCS + Citalopram + Rehabilitation (Experimental): * Real tDCS, 2 mA for 20 mins per session, 10 sessions within 2 weeks
  * Citalopram 10mg oral intake daily for 3 months, since 2 weeks before tDCS
  Interventions: Device: tDCS; Drug: Citalopram; Behavioral: Rehabilitation
- Sham tDCS + Citalopram + Rehabilitation (Sham Comparator): * Sham tDCS, ramped up over 10 seconds and then reduced to 0mA, 10 sessions within 2 weeks
  * Citalopram 10mg oral intake daily for 3 months, since 2 weeks before tDCS
  Interventions: Drug: Citalopram; Behavioral: Rehabilitation
- Real tDCS + Placebo + Rehabilitation (Placebo Comparator): * Real tDCS, 2 mA for 20 mins per session, 10 sessions within 2 weeks
  * Placebo oral intake daily for 3 months, since 2 weeks before tDCS
  Interventions: Device: tDCS; Behavioral: Rehabilitation
- Sham tDCS + Placebo + Rehabilitation (Placebo Comparator): * Sham tDCS, ramped up over 10 seconds and then reduced to 0mA, 10 sessions within 2 weeks
  * Placebo oral intake daily for 3 months, since 2 weeks before tDCS
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Device: tDCS — dual tDCS with ipsilesional primary motor cortex (M1) anodal stimulation and contralesional M1 cathodal stimulation, 2 weeks after SSRI treatment
  Arms: Real tDCS + Citalopram + Rehabilitation; Real tDCS + Placebo + Rehabilitation
Drug: Citalopram — total 3 months, since 2-4 weeks after stroke
  Arms: Real tDCS + Citalopram + Rehabilitation; Sham tDCS + Citalopram + Rehabilitation
Behavioral: Rehabilitation — hospitalized rehabilitation, 3 hours daily

SUMMARY:
Post-stroke motor recovery is compelling but limited. Current rehabilitation has less impacts on the plateau that spontaneous biological recovery could be expected. The advances in non-invasive neuromodulation and neurophysiological characterization of critical motor recovery period enable breaking the proportional recovery limitation. Our pilot studies demonstrated the safety and responsiveness of combing dual transcranial direct current stimulation (tDCS) and motor training in subacute stroke patients. There is also strong evidence that selective serotonin reuptake inhibitors (SSRIs) can substantially increase the effects of tDCS and improve motor function after stroke, even in the absence of depression. This proposal aims to prove the potential of combining of tDCS and the commonly used SSRI citalopram to improve response to a daily motor training intervention in acute stroke patients (Co-STARS trial).

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled study in 80 patients with first-ever, unilateral, subcortical ischemic stroke 0.5-4 weeks after stroke onset with moderate to severe hemiparesis. Participants were randomized into four groups underwent either real dual tDCS [ipsilesional primary motor cortex (M1) anodal stimulation and contralesional M1 cathodal stimulation; 2 mA for 20 mins; 10 sessions within 2 weeks] with citalopram or placebo, or sham stimulation with citalopram or placebo. All will receive concurrent hospitalized intensive rehabilitation of 2 daily sessions of 90-minute physiotherapy. Action reach am test (ARAT), Fugl-Meyer Assessment (FMA), multimodality MRI and EEG will be measured at baseline and after 2 weeks' tDCS modulation. The primary outcome is the ARAT at 3 months after intervention. The combination of tDCS and a SSRI will be expected to improve response to motor training more effectively than either intervention alone. The enhanced responsiveness will be correlated or predicted by biomarkers from multimodality MRI or EEG.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-80;
* first-onset stroke
* brain image confirmed unilateral subcortical infarction
* moderate to severe upper-limb impairment (SAFE score <8).
* 3 days to 4 weeks after stroke onset
* stable medical condition

Exclusion Criteria:

* metal implants, such as electrodes or pacemaker
* epilepsy history or active spikes from EEG recording
* major depression or taking psychoactive drugs
* alcoholism or drug abuse history
* combined with other severe neurological or psychiatric diagnoses
* pregnancy or breastfeeding;
* other contraindications to brain MRI, such as severe claustrophobia
* intolerance to electrical stimulation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Motor scores 3 months after intervention | 3 months after intervention
  Motor scores include Action research arm test (0-66, higher scores mean a better outcome) and Fugl-Meyer Assessment (0-54, higher scores mean a better outcome)